CLINICAL TRIAL: NCT02872272
Title: Amikacin Pharmacokinetic Profile in Plasma and Tissue After an Administration Using Impregnated Dressings in Burned Patient Population
Acronym: AMIKACINE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough participants to include
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-09; 2015-003972-64 (EudraCT Number)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Burn Patients
MeSH Terms: interventions — Therapeutics; Amikacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with Amikacin (Experimental): Dressing impregnated by administration of amikacin
  Interventions: Drug: Treatment with Amikacin

INTERVENTIONS:
Drug: Treatment with Amikacin — Aminoglycosides. Blood sampling for pharmacokinetic evaluation

SUMMARY:
The loss of skin barrier function after burn causes increased susceptibility to infections, which are the leading cause of morbidity and mortality in burn patients. Topical antibiotics are one part of the therapeutic arsenal available to treat these infections. Pseudomonas aeruginosa and Staphylococcus aureus are the two major colonizing agents found in this population of patients.

The use of dressings impregnated with amikacin is a common practice. Actually, there are no available data on local and systemic effects with this antibiotic. The study of tissue and plasma pharmacokinetics of amikacin is therefore very important to secure and optimize this singular use of amikacin and improve the care of burn patients.

The objective of the study is to describe the plasma and tissue pharmacokinetics of amikacin after dermal administration and impregnated dressing to estimate the pharmacokinetic parameters and their variability in a burned population.

Secondary objectives are to assess on the one hand the relationship between the effectiveness of treatment and the concentration of antibiotic at the site of tissue infection, and on the other hand to assess the relationship between plasma concentration and the toxicity found of this treatment. We would like also to note the efficacy of the antibiotic treatment in terms of: need for repeat surgery (new skin graft), healing time and hospital length of stay.

Blood samples and skin biopsies will be made for each patient to day 3 and day 7 after the start of treatment.

The knowledge about the tissue concentrations obtained and a possible systemic absorption will then provide additional safety data and optimize the conditions of use of these dressings (dosage, frequency of administration) for effective treatment and safe.

ELIGIBILITY:
Inclusion Criteria:

- Skin infection of burn (whatever the surface, depth or location) supported by percutaneous administration of amikacin Age greater than 18 years Patient can be under guardianship or trusteeship Patient may present with cognitive impairment Patients receiving social coverage Patient who understood the objectives of the study, agreeing to participate in the study and who signed informed consent (or for which a trustee or guardian signed an informed consent if necessary) Patient mastering the French language

Exclusion Criteria:

minor patient or pregnant or lactating deprived of liberty patient Patient does not have insurance coverage Patient does not agreeing to participate in the study Patient allergic to amikacin or other antibiotic aminoglycosides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Determination of amikacin concentration | 24 months
  Concentration of amikacin in nanograms per milliliter. Circulating amikacin will be quantified by chromatographic high-performance technology

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No